CLINICAL TRIAL: NCT06396975
Title: Comparison of Short-term Outcomes of Robotic and Laparoscopic Surgery in Patients With Different Body Mass Index for Mid and Low Rectal Cancer
Status: Completed | Type: Observational
Sponsor: Daorong Wang (Other)
Responsible Party: Sponsor-Investigator, Daorong Wang, Dr, Northern Jiangsu People's Hospital
Organization: Northern Jiangsu People's Hospital (Other)
Other Study IDs: Northjiangsu020
Record Dates: First submitted 2024-04-29; First posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Robotic Surgical Procedures

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- laparoscopic surgery
  Interventions: Procedure: robotic surgery
- robotic surgery
  Interventions: Procedure: robotic surgery

INTERVENTIONS:
Procedure: robotic surgery — robotic surgery

SUMMARY:
Numerous comparison studies on the outcomes of robotic and laparoscopic surgery in the treatment of rectal cancer have been undertaken and reported. But there aren't many studies that compare the safety and effectiveness of the two surgery procedures used to treat people with mid and low rectal cancer who have different body mass indexes (BMIs). This study was done to organize the clinical data we had at our hospital so we could compare the perioperative effectiveness of two minimally invasive approaches for people with different BMIs.

ELIGIBILITY:
Inclusion Criteria:

The inclusion decision was made based on the following criteria: the results of the preoperative evaluation revealed the existence of adenocarcinoma in the middle to lower rectum (less than 10 centimeters distant from the anal edge); received a drastic operation that might have been laparoscopic or robotic and was based on the principle of TME; distant metastases that are non-conformist or heteroclinic, and there are no additional malignant tumors present at the same time as the operation.

Exclusion Criteria:

a high tumor location that was more than 10 centimeters away from the anal margin; surgery was unsuccessful in completing anal preservation due to invasion of the external anal sphincter; cancerous obstruction or perforation; severe cardiopulmonary dysfunction classified as stage IV according to the ASA score; and poor preoperative anal function; any resection that is performed in combination, rather than being a R0 resection.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The clinical records of patients who had laparoscopic or robotic proctectomy at Northern Jiangsu People's Hospital between December 2019 and August 2023 were analyzed in order to conduct research utilizing a retrospective research technique.
Sampling Method: Non-Probability Sample
Enrollment: 1413 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-04-29 (Actual); Study Completion 2024-04-29 (Actual)

PRIMARY OUTCOMES:
Oncological outcomes | 2019-2023
  Oncological outcomes
the frequency of complications | 2019-2023
  the frequency of complications

CONTACTS AND LOCATIONS:
Locations (1):
- Northern Jiangsu People's Hospital, Yangzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No